CLINICAL TRIAL: NCT01250106
Title: Phase I Study of Probiotics as a Novel Approach to Modulate Gut Hormone Secretion and Risk Factors of Type 2 Diabetes and Complications
Brief Title: Probiotics as a Novel Approach to Modulate Gut Hormone Secretion and Risk Factors of Type 2 Diabetes and Complications
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: German Diabetes Center (Other)
Collaborators: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Schloot, Nanette C., German Diabetes Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Probiotic-01
Record Dates: First submitted 2010-11-24; First posted 2010-11-30 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: probiotics; prevention; dietary intervention; insulin resistance; obesity; type 2 diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic capsule (Experimental)
  Interventions: Dietary Supplement: Lactobacillus reuteri
- placebo capsule (Placebo Comparator)
  Interventions: Dietary Supplement: Lactobacillus reuteri

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri — twice daily

SUMMARY:
The investigators aim to test the hypothesis that Lactobacillus Reuteri-enriched microbiota improves insulin sensitivity and glucose tolerance in obese healthy and obese type 2 diabetes patients by improving gut hormone secretion and compare these findings to healthy lean subjects.

DETAILED DESCRIPTION:
Prediabetes and diabetes are accompanied by insufficient gut hormone release, insulin resistance, insufficient insulin secretory capacity and low grade systemic inflammation. Results of recent animal experiments suggest that ingestion of probiotics not only influences gut microbiota composition and intestinal permeability but also secretion of GLP-2 as well as insulin resistance, components of metabolic syndrome and diabetes development. GLP-2 secretion has been suggested to be a key mediator of probiotic effects mediating decreased intestine permeability through binding to intestinal GLP2 receptor in animal studies. Insulinotropic GLP-1, which is reduced in patients with type 2 diabetes, has also been described to be influenced by gut microbiota composition. We aim to test the hypothesis that Lactobacillus Reuteri-enriched microbiota improves insulin sensitivity and glucose tolerance in obese healthy and obese type 2 diabetes patients by improving gut hormone secretion. In a prospective, double-blinded, placebo controlled randomized 10 weeks trial we aim to investigate metabolic and immunological changes related to modified gut microbiota by analysing (1) gut hormone secretion, (2) insulin sensitivity and glucose tolerance, and (3) systemic LPS concentrations and immune status.

ELIGIBILITY:
Inclusion Criteria:

* Obese subjects: age 40 - 65 years, obesity (BMI 30-45 kg/m2), non-smoking, absence of gastrointestinal disease, willingness to abstain from intake of fermented milk products over a study period of 8 weeks.
* Healthy control subjects: non-obese (BMI 19-25 kg/m2), non-diabetic subjects, matched for age and sex, non-smoking, absence of gastrointestinal disease, willingness to abstain from intake of fermented milk products over a study period of 8 weeks.

Exclusion Criteria:

* pregnancy, cancer, chronic diseases, antibiotic therapy, competitive athletes.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Insulin resistance | 8 weeks

SECONDARY OUTCOMES:
gut hormones (GLP-1, GLP-2, GIP) | 8 and 10 weeks
insulin secretion | 8 and 10 weeks
measurement of cytokines to define the immune status | 8 and 10 weeks
  measurement and analysis of proinflammatory cytokines (Interleukin (IL)-6, tumor necrosis factor (TNF)-α, IL-1ß, Macropahge inflammatory protein (MIP)-1ß) and regulatory cytokines (IL-10, transforming growth factor (TGF)-ß, IL1ra) from peripheral blood samples collected during this trial
body weight | 8 and 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nanette C Schloot, Priv.-Doz. MD, Principal Investigator — German Diabetes Center, Duesseldorf
Locations (1):
- German Diabetes Center, Düsseldorf, Duesseldorf, Germany

REFERENCES:
- [Derived] Simon MC, Strassburger K, Nowotny B, Kolb H, Nowotny P, Burkart V, Zivehe F, Hwang JH, Stehle P, Pacini G, Hartmann B, Holst JJ, MacKenzie C, Bindels LB, Martinez I, Walter J, Henrich B, Schloot NC, Roden M. Intake of Lactobacillus reuteri improves incretin and insulin secretion in glucose-tolerant humans: a proof of concept. Diabetes Care. 2015 Oct;38(10):1827-34. doi: 10.2337/dc14-2690. Epub 2015 Jun 17. PMID 26084343